CLINICAL TRIAL: NCT06476236
Title: M4C Nutraceutical Intervention Human Health Effects Pilot
Acronym: M4C Pilot
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Concordia University Wisconsin (Other)
Responsible Party: Principal Investigator, Joseph McGraw, Professor, Concordia University Wisconsin
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: IRB-FY24-293
Record Dates: First submitted 2024-06-05; First posted 2024-06-26 (Actual); Last update posted 2024-06-26 (Actual); Status verified 2024-06

CONDITIONS: General Health and Wellness; Energy and Vitality; Cognitive Function and Mental Health; Weight Management; Digestive Health; Exercise Tolerance; Cardiovascular Health; Bone and Joint Health; Skin, Hair, and Nail Health; Immune Support; Sports Performance and Recovery; Sleep and Relaxation; Obesity; Anti Inflammatory
Keywords: General Health and Wellness; Energy and Vitality; Cognitive Function and Mental Health; Weight Management; Digestive Health; Exercise Tolerance; Cardiovascular Health; Bone and Joint Health; Skin, Hair, and Nail Health; Immune Support; Sports Performance and Recovery; Sleep and relaxation; Obesity; anti inflammatory
MeSH Terms: conditions — Psychological Well-Being; Obesity

STUDY DESIGN:
Intervention Model Description: Open label single arm intervention pilot
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- M4C Treatment (Experimental): Single arm study with nutraceutical M4C treatment. Proprietary blend of amino acids, fatty acids, vitamins, and minerals. 1 tbsp in 12 oz of water with two algae oil capsules taken by mouth one to two times daily.
  Interventions: Dietary Supplement: M4C

INTERVENTIONS:
Dietary Supplement: M4C — Nutraceutical designed to enhance novel metabolic pathway activity.

SUMMARY:
This 3 month pilot study will be an unblinded, convenience sampling, nutraceutical intervention trial. Twenty fasted subjects will undergo a baseline health assessment via a questionnaire, baseline clinical chemistries, blood lipids, dexa and impedence testing (to identify bone mineral density and body muscle/fat/water composition), and metabolite/novel biomarker testing through whole capillary blood, saliva, and urine collections. Assessments will be repeated every month (3 times after initial assessment) to cover a 3 month period. All measurements from each visit will be compared with baseline using paired t-tests or Chi square testing depending on variable. Power analyses are not included due to the pilot nature of the study. This pilot study will provide the necessary variability estimates for future trials.

DETAILED DESCRIPTION:
The purpose of this study is to explore potential positive human health effects of a proprietary nutraceutical formulation known as M4C. The impetus for M4C came from Dr. McGraw's attempt to alleviate the chronic inflammation a family member was experiencing through a non-invasive, natural, nutraceutical approach. Anecdotal findings of M4C show an antiinflammatory effect (observed in the presence of inflammatory conditions and after traumatic injury such as a sprain or fall), improved metabolic, gastrointestinal, and mental health, as well as enhanced exercise response and recovery. In this study the investigators will examine whether supplementation with M4C is associated with any changes in lipids, clinical chemistries, body composition, questionnaire covariates, metabolites/novel suspected lipopeptides, hemoglobin A1C, or bone mineral density.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults

Exclusion Criteria:

* amputation
* blood clotting disorder
* metal implants or implanted electrical device(s)
* known acute or chronic illness; gastrointestinal, cardiac, pulmonary, liver, or kidney abnormalities, uncontrolled hypertension
* inability to fast i.e. low blood sugar
* pregnant or may be pregnant during the course of the study
* amino acid metabolizing disorder i.e. phenylketonuria
* severe edema
* did not pass screening criteria as determined by MRI facility
* allergies/intolerance to any nutraceutical ingredients: amino acids, vitamins, minerals, tapioca starch, sunflower lecithin, stevia, limes or fatty acids like docosahexaenoic acid

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-06-17 (Estimated); Primary Completion 2025-06-17 (Estimated); Study Completion 2025-06-17 (Estimated)

PRIMARY OUTCOMES:
Body composition | 3 months
  Dexa scan for bone mineral density
Body composition | 3 months
  Dexa scan for body fat distribution
Body composition | 3 months
  Dexa scan for body muscle distribution
Hemoglobin A1C | 3 months
  measured glycated hemoglobin via whole capillary blood
Resting Systolic blood pressure | Monthly for 3 months
  measured via Omron Platinum digital upper arm blood pressure monitor
Resting Diastolic blood pressure | Monthly for 3 months
  measured via Omron Platinum digital upper arm blood pressure monitor
Resting Pulse | Monthly for 3 months
  measured via Omron Platinum digital upper arm blood pressure monitor
Blood lipids | Monthly for 3 months
  measured via blood lipid analyzer from whole capillary blood
Anxiety | Monthly for 3 months
  Measured via Generalized Anxiety Disorder (GAD-7) questionnaire Scoring as follows 0-4: No anxiety, 5-9:Mild anxiety, 10-14:Moderate anxiety, 15-21: Severe anxiety
General Mental Health | Monthly for 3 months
  User rating as follows: Excellent, Very good, Good, Fair, Poor
Chronic Pain | Monthly for 3 months
  Self reported chronic pain as follows: Self rated from 0-10 Zero is no pain, 10 is worst pain imaginable

SECONDARY OUTCOMES:
Saliva Melatonin and Cortisol | 3 months
  Concentrations of melatonin and cortisol in saliva (ng/ml) will be collected before bedtime and at rising. Sample melatonin and cortisol will be measured via High Performance liquid chromatography with mass spectrometry (HPLC MS/MS) as potential markers of stress state. Values will be assessed for conformance to reported reference ranges in the literature. Values outside the reference ranges will be considered positive for unhealthy stress response.

CONTACTS AND LOCATIONS:
Overall Officials: Tonya Bartoletti, Study Director — Concordia University of Wisconsin ORSP assistant director

IPD SHARING:
Plan to Share IPD: No